CLINICAL TRIAL: NCT04362566
Title: Randomized Trial of Bupivacaine as Adjuvant for Post-operative Pain in Mohs Micrographic Surgery
Brief Title: Bupivacaine for Post-operative Pain in Mohs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Pennsylvania (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Nicholas J Golda, Professor, Dermatology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022277
Record Dates: First submitted 2020-04-16; First posted 2020-04-27 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Pain, Postoperative; Narcotic Use
Keywords: local anesthetic
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Single-blind RCT
Who Masked: Participant
Masking Description: Patients will receive long acting local anesthetic or saline placebo postoperatively, they will be blinded to the arm they are in
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivicaine (Active Comparator): Scalp flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc, Ear flap or wedge repair: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Nose flap, 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc. Split volume between nose and donor site for melolabial interpolated flap Paramedian forehead flap: 5cc split between forehead donor site and nasal recipient site: 4cc forehead, 1cc nose Cartilage alar-batten graft (ear donor site) 1cc at auricular donor site in addition to bupivacaine used for nasal reconstruction, if any, that qualifies above Cheek Mustarde flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Lip flap, wedge repair, Abbe flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc
  Interventions: Drug: Bupivacaine
- Placebo saline (Placebo Comparator): Saline in the same volume as described above for bupivicaine
  Interventions: Other: Placebo Saline

INTERVENTIONS:
Drug: Bupivacaine — Scalp flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc, Ear flap or wedge repair: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Nose flap, 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc. Split volume between nose and donor site for melolabial interpolated flap Paramedian forehead flap: 5cc split between forehead donor site and nasal recipient site: 4cc forehead, 1cc nose Cartilage alar-batten graft (ear donor site) 1cc at auricular donor site in addition to bupivacaine used for nasal reconstruction, if any, that qualifies above Cheek Mustarde flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Lip flap, wedge repair, Abbe flap: 2.5cc bupivacaine for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc
  Arms: Bupivicaine
Other: Placebo Saline — Scalp flap: 2.5cc salinefor 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc, Ear flap or wedge repair: 2.5cc saline for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Nose flap, 2.5cc saline for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc. Split volume between nose and donor site for melolabial interpolated flap Paramedian forehead flap: 5cc split between forehead donor site and nasal recipient site: 4cc forehead, 1cc nose Cartilage alar-batten graft (ear donor site) 1cc at auricular donor site in addition to saline used for nasal reconstruction, if any, that qualifies above Cheek Mustarde flap: 2.5cc saline for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc Lip flap, wedge repair, Abbe flap: 2.5cc saline for 0-10cm2, additional 1cc for each additional 10cm2 up to max 5cc
  Arms: Placebo saline

SUMMARY:
Mohs micrographic surgery (MMS) is regarded as the gold standard for the treatment of high-risk nonmelanoma skin cancer (NMSC). Pain after MMS peaks on the day of surgery and slowly decreases thereafter. The most common post-operative analgesics include acetaminophen, ibuprofen and narcotics. Lidocaine is the most commonly used anesthetic in MMS, but bupivacaine has been shown in other surgical specialties to be an effective adjuvant to reduce post-operative pain and opioid use when injected locally in the immediate postoperative period. Bupivacaine has also been shown to reduce intra-operative pain during MMS. The investigators plan a single-blinded prospective, randomized, controlled trial to determine if post-operative wound infiltration of bupivacaine versus normal saline improves post-operative pain and decreases need for post-operative pain medications including both narcotic and nonnarcotic analgesics.

DETAILED DESCRIPTION:
Mohs micrographic surgery (MMS) is the first-line treatment for high-risk nonmelanoma skin cancer (NMSC) and is increasingly used for melanoma and other cutaneous neoplasms. The surgical technique involves multiple stages of surgery followed by reconstruction and is typically performed under local anesthesia in the office setting in one day.

MMS is generally well tolerated, but post-operative pain is common. Pain peaks on the day of surgery and slowly declines in subsequent days. Risk factors for increased pain may include flap or graft repair type, location on scalp, lip, nose, or ear, younger age, and increased number of lesions treated. Post-operative pain medication is not standardized in dermatological surgery, but often includes non-narcotic analgesics including acetaminophen and ibuprofen, and less commonly narcotic analgesics such as tramadol and oxycodone. Given the current national trend to reduce opioid use, a multimodal approach to pain management has been adopted by many surgical specialties to optimize analgesia perioperatively.

The most commonly used anesthetic in MMS is local subcutaneous infiltration of lidocaine 0.5 - 2% with 1:100,000 - 1:200,000 epinephrine. Lidocaine is quick-acting, can be buffered to reduce injection pain, and is well tolerated, but the duration of action is only two hours, making it less effective for post-operative pain. Bupivacaine with epinephrine has a longer duration of action compared to lidocaine (up to four hours), but it is rarely used alone due to slower onset of action and more painful injection compared with lidocaine. Bupivacaine is used in many other surgical specialties, including general, plastic, and orthopedic surgery, as a peri-operative adjuvant and has been shown to reduce post-operative opioid use. It is generally well tolerated, carrying a class-effect risk of cardiac toxicity in high doses as does lidocaine, but has been shown to be safe in dermatologic surgery when used for wound infiltration. A newer formulation of liposomal bupivacaine has been shown to be even longer lasting and safer, with pain control up to 72 hours and no reported cardiac toxicity. In addition, a recent study has showed subcutaneous infiltration of bupivacaine with epinephrine to be an effective intra-operative pain adjuvant during MMS compared to lidocaine alone.

Pain control post-operatively in MMS may be optimized by including bupivacaine injections at the end of the surgical procedure given its long-lasting anesthetic effects. There are currently no studies addressing the use of bupivacaine as an adjuvant to control post-operative pain during MMS. The investogators propose a prospective randomized controlled trial to evaluate the effectiveness of bupivacaine injection at the conclusion of surgery for reducing post-operative pain and analgesic use.

ELIGIBILITY:
Inclusion Criteria:

* a. Adult (18 years or older) patients being treated with Mohs micrographic surgery will be included in this study.

  b. Surgical procedure must include one of the following:
  1. Scalp rotation/transposition/advancement flap
  2. Ear rotation/transposition/advancement/interpolation flap or wedge repair
  3. Nose rotation/transposition/advancement/interpolation flap, cartilage alar-batten graft (ear donor site)
  4. Cheek Mustarde flap
  5. Lip rotation/transposition/advancement flap, wedge repair, Abbe flap

     Exclusion Criteria:
* c. Patients must not

  1. be pregnant or breastfeeding
  2. be taking scheduled narcotic medications
  3. use narcotics as a drug of abuse
  4. have an allergy to bupivacaine or other amide anesthetics
  5. have a contraindication to tramadol
  6. have been given narcotic pain medications during the Mohs procedure or subsequent reconstruction
  7. have multiple surgical sites treated on the same day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pain control | 24 hours
  Determination if bupivacaine injection postoperatively in clinical scenarios where higher postoperative pain is expected (see protocol) changes the need for narcotic medication (using a binary Yes or No measure) during first 24 hours post-surgery

SECONDARY OUTCOMES:
48 hour pain control 1-10 scale | 48 hours
  Postoperative pain levels (1-10 scale) during 48 hours following surgery in the intervention and control groups
48 hour pain control drug type used if any | 48 hours
  48 hour pain control drug type (narcotic versus nonnarcotic versus none) in the intervention and control groups
48 hour pain control drug amount used if any | 48 hours
  Determination of the amount (number of doses) of various pain control drugs (narcotic versus nonnarcotic versus none) needed during 48 hours following operation and calculating if there is a difference between the intervention and control groups
Adverse effects | 48 hours
  Documenting adverse effects, if any, from long-acting anesthetic that are different from the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Golda, MD, Principal Investigator — University of Missouri School of Medicine
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Patient data will be submitted from University of Pennsylvania and Columbia university to the University of Missouri primary research group for statistical analysis. The IPD will not be shared outside of this research team.

REFERENCES:
- [Background] Tolkachjov SN, Brodland DG, Coldiron BM, Fazio MJ, Hruza GJ, Roenigk RK, Rogers HW, Zitelli JA, Winchester DS, Harmon CB. Understanding Mohs Micrographic Surgery: A Review and Practical Guide for the Nondermatologist. Mayo Clin Proc. 2017 Aug;92(8):1261-1271. doi: 10.1016/j.mayocp.2017.04.009. PMID 28778259
- [Background] Saco M, Golda N. Postoperative Pain Management in Dermatologic Surgery: A Systematic Review. Dermatol Clin. 2019 Jul;37(3):341-348. doi: 10.1016/j.det.2019.03.004. Epub 2019 Apr 16. PMID 31084728
- [Background] Saco M, Golda N. Optimal timing of postoperative pharmacologic pain control in Mohs micrographic surgery: A prospective cohort study. J Am Acad Dermatol. 2020 Feb;82(2):495-497. doi: 10.1016/j.jaad.2019.07.077. Epub 2019 Jul 30. No abstract available. PMID 31374303
- [Background] Roy CF, Azzi AJ, Davison P. A Review of Wound Infusion With Local Anesthetics in Plastic Surgery. Ann Plast Surg. 2019 Dec;83(6):e110-e117. doi: 10.1097/SAP.0000000000001916. PMID 31192870
- [Background] Dasta J, Ramamoorthy S, Patou G, Sinatra R. Bupivacaine liposome injectable suspension compared with bupivacaine HCl for the reduction of opioid burden in the postsurgical setting. Curr Med Res Opin. 2012 Oct;28(10):1609-15. doi: 10.1185/03007995.2012.721760. Epub 2012 Sep 3. PMID 22900785
- [Background] Chen P, Smith H, Vinciullo C. Bupivacaine as an Adjunct to Lidocaine in Mohs Micrographic Surgery: A Prospective Randomized Controlled Trial. Dermatol Surg. 2018 May;44(5):607-610. doi: 10.1097/DSS.0000000000001385. PMID 29140864
- [Background] Merritt BG, Lee NY, Brodland DG, Zitelli JA, Cook J. The safety of Mohs surgery: a prospective multicenter cohort study. J Am Acad Dermatol. 2012 Dec;67(6):1302-9. doi: 10.1016/j.jaad.2012.05.041. Epub 2012 Aug 11. PMID 22892283
- [Background] Limthongkul B, Samie F, Humphreys TR. Assessment of postoperative pain after Mohs micrographic surgery. Dermatol Surg. 2013 Jun;39(6):857-63. doi: 10.1111/dsu.12166. Epub 2013 Mar 6. PMID 23464845
- [Background] Firoz BF, Goldberg LH, Arnon O, Mamelak AJ. An analysis of pain and analgesia after Mohs micrographic surgery. J Am Acad Dermatol. 2010 Jul;63(1):79-86. doi: 10.1016/j.jaad.2009.10.049. PMID 20542176
- [Background] Sniezek PJ, Brodland DG, Zitelli JA. A randomized controlled trial comparing acetaminophen, acetaminophen and ibuprofen, and acetaminophen and codeine for postoperative pain relief after Mohs surgery and cutaneous reconstruction. Dermatol Surg. 2011 Jul;37(7):1007-13. doi: 10.1111/j.1524-4725.2011.02022.x. Epub 2011 May 11. PMID 21561527
- [Background] Evans T, Nicholas TA, Sutton AV, Wysong A. How We Do It: Postoperative Pain Control in Mohs Micrographic Surgery. Dermatol Surg. 2021 Feb 1;47(2):280-282. doi: 10.1097/DSS.0000000000002279. No abstract available. PMID 31809346
- [Background] Lovich-Sapola J, Smith CE, Brandt CP. Postoperative pain control. Surg Clin North Am. 2015 Apr;95(2):301-18. doi: 10.1016/j.suc.2014.10.002. Epub 2015 Jan 24. PMID 25814108
- [Background] Park KK, Sharon VR. A Review of Local Anesthetics: Minimizing Risk and Side Effects in Cutaneous Surgery. Dermatol Surg. 2017 Feb;43(2):173-187. doi: 10.1097/DSS.0000000000000887. PMID 27608208
- [Background] Kouba DJ, LoPiccolo MC, Alam M, Bordeaux JS, Cohen B, Hanke CW, Jellinek N, Maibach HI, Tanner JW, Vashi N, Gross KG, Adamson T, Begolka WS, Moyano JV. Guidelines for the use of local anesthesia in office-based dermatologic surgery. J Am Acad Dermatol. 2016 Jun;74(6):1201-19. doi: 10.1016/j.jaad.2016.01.022. Epub 2016 Mar 4. PMID 26951939
- [Background] Sorenson E, Chesnut C. Liposomal Bupivacaine: A Review and Applications to Dermatologic Surgery. Dermatol Surg. 2019 Jan;45(1):68-73. doi: 10.1097/DSS.0000000000001628. No abstract available. PMID 30148736
- See also: Bupivicaine drug insert — https://www.accessdata.fda.gov/drugsatfda_docs/label/2010/071168s020lbl.pdf